CLINICAL TRIAL: NCT05367349
Title: Optimising Screening for Early Disease Detection in Familial Pulmonary Fibrosis
Acronym: FLORIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Antonius Hospital (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Jan C. Grutters, MD, Prof. Dr., St. Antonius Hospital
Other Study IDs: NL75303.100.20
Record Dates: First submitted 2022-03-28; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Fibrosis Idiopathic Familial
Keywords: Pulmonary Fibrosis; Familial; Screening; Asymptomatic; Family members; First-degree
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators will store the following tubes:
  One CPT tube / One EDTA tube / One lithium-heparin tube, each divided in three aliquots / Two serum tubes, each divided in three aliquots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study the prognostic value of the current screening parameters for familial pulmonary fibrosis (FPF) will be investigated by looking at the screenings of 200 first-degree relatives of patients with FPF.

Also insight in the natural history of early FPF, and the necessary interval between screenings visits will be investigated.

DETAILED DESCRIPTION:
Familial pulmonary fibrosis (FPF) is a fatal lung disease that is often not diagnosed until a significant portion of the lung function is lost. Median survival after diagnosis is 3 to 5 years. As treatment can only slow down lung function decline, early disease detection is essential to provide timely therapeutic support. As first-degree relatives of patients with FPF are at high risk of developing pulmonary fibrosis as well, a screening protocol has been put in place. However, the value of current screening parameters to detect early asymptomatic disease as well as the optimal interval between screening appointments are unknown. A prospective study into the prognostic value of these screening markers in the target population and the appropriate clinical setting is needed to develop an evidence-based screening protocol. There will be an emphasis on easily operable parameters that may allow for redirection of (part of the) screening activities to the general practice in the future.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic first-degree relative of patients with familial pulmonary fibrosis (FPF)

Exclusion Criteria:

* A previous diagnosis of interstitial lung disease (ILD)
* Minors (aged <18 years)
* Pregnant

Note: woman who are pregnant at the start of the study or at the time of the HRCT are not allowed to participate. If a participant gets pregnant at a later stage during the study, she will not be excluded from the study. To be able to account for a potential effect of pregnancy during data analysis, female participants can be asked if they are pregnant at every visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymptomatic first-degree relatives of patients with FPF are invited to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2025-06-16 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Characteristics of participants | Baseline
  Difference in age, sex, body weight, smoking history and comorbidities between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Forced Vital Capacity (FVC) | Baseline
  Difference in forced vital capacity (FVC) between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Haemoglobulin-corrected carbon monoxide diffusing capacity (DLCOc) | Baseline
  Difference in haemoglobulin-corrected carbon monoxide diffusing capacity (DLCOc) between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Total lung capacity (TLC) | Baseline
  Difference in total lung capacity (TLC) between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Biomarker levels | Baseline
  Difference in Krebs von den Lungen 6 (KL6), chemokine (C-C motif) ligand 18 (CCL18), surfactant protein-D (SP-D), matrix metalloproteinase 7 (MMP7) between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Oxygen saturation in 6-minute walk test (6MWT) | Baseline
  Difference in oxygen saturation (rest in %), oxygen saturation (after 6MWT in %), oxygen saturation (nadir in %) and oxygen saturation (difference between rest and nadir in %) (all continuous variables) between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Distance (meters) in 6-minute walk test (6MWT) | Baseline
  Difference in distance covered (in meters) between the group with ILD changes and the group without ILD changes present on enrollment HRCT
MUC5B genotype | Baseline
  Difference in MUC5B genotype (all discrete variables) between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Patient reported cough score | Baseline
  Difference in visual analogue scale (VAS) for cough (scores between 0-100, with 100 being the worst) between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Patient reported dyspnea score | Baseline
  Difference in medical research council (MRC) (scores between 0-5, with 5 being the worst) between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Clubbing | Baseline
  Difference in presence of digital clubbing between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Crackles | Baseline
  Difference in inspiratory crackles during lung auscultation between the group with ILD changes and the group without ILD changes present on enrollment HRCT

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | 2 years
  Difference in forced vital capacity (FVC) over the course of 2 years in the subjects with presence of ILD changes on enrollment HRCT and also between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Haemoglobulin-corrected carbon monoxide diffusing capacity (DLCOc) | 2 years
  Difference in haemoglobulin-corrected carbon monoxide diffusing capacity (DLCOc) over the course of 2 years in the subjects with presence of ILD changes on enrollment HRCT and also between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Total lung capacity (TLC) | 2 years
  Difference in total lung capacity (TLC) over the course of 2 years in the subjects with presence of ILD changes on enrollment HRCT and also between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Biomarker levels | 2 years
  Difference in KL6, CCL18, SP-D and MMP7 over the course of 2 years in the subjects with presence of ILD changes on enrollment HRCT and also between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Genotype | 2 years
  Difference in MUC5B genotype over the course of 2 years in the subjects with presence of ILD changes on enrollment HRCT and also between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Oxygen saturation in 6-minute walk test (6MWT) | 2 years
  Difference in oxygen saturation (rest in %), oxygen saturation (after 6MWT in %), oxygen saturation (nadir in %) and oxygen saturation (difference between rest and nadir in %) (all continuous variables) over the course of 2 years in the subjects with presence of ILD changes on enrollment HRCT and also between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Distance (meters) in 6-minute walk test (6MWT) | 2 years
  Difference in distance covered (in meters) over the course of 2 years in the subjects with presence of ILD changes on enrollment HRCT and also between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Patient reported cough score | 2 years
  Difference in visual analogue scale (VAS) for cough (scores between 0-100, with 100 being the worst) over the course of 2 years in the subjects with presence of ILD changes on enrollment HRCT and also between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Patient reported dyspnea score | 2 years
  Difference in medical research council (MRC) (scores between 0-5, with 5 being the worst) over the course of 2 years in the subjects with presence of ILD changes on enrollment HRCT and also between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Digital clubbing | 2 years
  Difference in presence of digital clubbing over the course of 2 years in the subjects with presence of ILD changes on enrollment HRCT and also between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Crackles | 2 years
  Difference in inspiratory crackles during lung auscultation over the course of 2 years in the subjects with presence of ILD changes on enrollment HRCT and also between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Patient reported fatigue | 2 years
  Difference in fatigue assessment scale (FAS) (scores range from 10-50, with 50 being the worst) over the course of 2 years in the subjects with presence of ILD changes on enrollment HRCT and also between the group with ILD changes and the group without ILD changes present on enrollment HRCT
Patient reported health status | 2 years
  Difference in EuroQol 5D-5L (EQ-5D-5L) (comprises of a score in five levels, level 1-5 with 5 being the worst, and a visual analoque scale ranging from 0-100 with 100 being the best) and the over the course of 2 years in the subjects with presence of ILD changes on enrollment HRCT and also between the group with ILD changes and the group without ILD changes present on enrollment HRCT

OTHER OUTCOMES:
Relatedness | Baseline
  In case multiple members of the same family are included in the study
Blood count | 2 years
  Blood count (Consisting of; hemoglobin (mmol/l), erythrocytes (x10^12/l), mean corpuscular volume (fl), red cell distribution width (%), thrombocytes (x10^9/l), leukocytes (x10^9/l)) as an exploratory measurement in the subjects with presence of ILD changes on enrollment HRCT and the difference between bloodcount in the subjects with presence of ILD changes on enrollment HRCT and the group without ILD changes present on enrollment HRCT
Creatinin | 2 years
  creatinin (umol/l) as an exploratory measurement in the subjects with presence of ILD changes on enrollment HRCT and the difference between creatinin in the subjects with presence of ILD changes on enrollment HRCT and the group without ILD changes present on enrollment HRCT
Liver function tests | 2 years
  Liver function tests (consisting of: ASAT (U/l), ALAT (U/l), alkaline phosphatase (U/l), Gamma-glutamyl transpeptidase (U/l)) as an exploratory measurement in the subjects with presence of ILD changes on enrollment HRCT and the difference between these liver function tests in the subjects with presence of ILD changes on enrollment HRCT and the group without ILD changes present on enrollment HRCT
Total bilirubin | 2 years
  Total bilirubin (umol/l) as an exploratory measurement in the subjects with presence of ILD changes on enrollment HRCT and the difference between total bilirubin in the subjects with presence of ILD changes on enrollment HRCT and the group without ILD changes present on enrollment HRCT
Additional blood based markers | 2 years
  Additional blood based markers as an exploratory measurement in the subjects with presence of ILD changes on enrollment HRCT and the difference between these blood based markers in the subjects with presence of ILD changes on enrollment HRCT and the group without ILD changes present on enrollment HRCT

CONTACTS AND LOCATIONS:
Locations (1):
- St Antonius Hospital, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data of patients is coded